CLINICAL TRIAL: NCT04280523
Title: TranspulmonarY Estrogen Gradient and Estrogen Receptors (TYEGER) in PAH
Acronym: TYEGER
Status: Withdrawn | Type: Observational
Why Stopped: The study was withdrawn, with no participants enrolled.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Eric Austin, Associate Professor of Pediatrics, Director Vanderbilt Pediatric PH Program, Vanderbilt University Medical Center
Other Study IDs: 191946
Record Dates: First submitted 2020-01-15; First posted 2020-02-21 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — 16-fluoroestradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- ESR-specific PET Scan: Specific Aim: To test the hypothesis that among PAH patients, higher lung ESR density associates with a more severe hemodynamic profile and worse 1 year outcomes.
  Study Design: Enroll 20 randomly selected subjects from each group (PAH vs. control)
  Interventions: Drug: ESR-specific PET scan

INTERVENTIONS:
Drug: ESR-specific PET scan — Lung ESR Density by PET: Investigators will use 18F-FES as an estrogen receptor (ESR)-specific PET tracer to determine lung ESR density. 18F-FES will be prepared according to published methods. Briefly, all subjects will be evaluated by PET imaging, using standardized protocols. Blood will be obtained just before FES injection to measure the endogenous estrogen level [estradiol (E2)], to rule out pregnancy in female patients, and some reserved for future studies of mechanism. Approximately 6 mCi (222 MBq) of 18F-FES will be administered intravenously over 1~2 minutes, with scanning initiated 1 hour after administration of the tracer. Emission scans will be performed of the chest. A multimodality computer platform (Syngo; Siemens) will be used for image review and manipulation.
  Other Names: [18F]FES

SUMMARY:
Pulmonary arterial hypertension (PAH) is a disease characterized by elevated pressures in the blood vessels of the lungs that is not caused by another disease processes. More specifically, it is defined by a mean pulmonary artery pressure > 25 mm Hg, a pulmonary vascular resistance > 3 Wood Units (WU), and a normal pulmonary capillary wedge pressure in the absence of other etiology of pulmonary hypertension. The underlying mechanism of the disease in still unknown, but marked changes to the small arteries in the lungs have been observed. These changes include thickening of vessel walls and clot formation -- making the vessels less capable of gas exchange. Currently, PAH therapies focus on dilating the "good" remaining vessels that haven't been altered by this disease process; however, this therapy does not cure the disease. Survival remains low despite progress.

There is growing human and experimental evidence supporting the concept that estrogens and estrogen receptors in the lungs are involved in the process that leads to PAH.

As mentioned above, no current therapies attack the cause of PAH; they only act to dilate remaining "good" vessels which can reduce the burden of the disease, but not cure it. Thus, there is a critical need for novel therapeutics, as recently highlighted by a National Institute of Health workshop on pulmonary vascular diseases which called for the exploration of novel therapeutic approaches. None of the current FDA-approved treatments for PAH target estrogen or estrogen receptors.

Despite the evidence supporting the concept that estrogens and estrogen receptors in the lungs contribute to PAH, no human studies investigate the estrogen level and the amount of estrogen receptors within the lungs of patients with PAH and their potential associations with current disease severity or 1 year outcomes including survival after 1 year, functional status, etc. Investigators hypothesize that a subset of PAH patients will have higher levels of estrogen and estrogen receptors in their lungs which would make them good candidates for novel therapies that block estrogen in hopes of halting the disease process.

Update 12/31/2024:

This record was updated to reflect the actual status of the research:

* The study was observational, as the 18F-FES PET was not an interventional procedure, but was planned to be used as an estrogen receptor (ESR)-specific PET tracer to determine lung ESR density.
* Zero participants were enrolled. Due to Covid-19, we utilized 66 serum samples from another study to test the hypothesis that among PAH patients, transpulmonary (TP) E2 gradient associates with a more severe hemodynamic profile and worse 1 year outcomes.

DETAILED DESCRIPTION:
The strongest established risk factor for the progressively fatal disease pulmonary arterial hypertension (PAH) is female sex (~3:1 female:male ratio). Investigators and others have found higher circulating estrogen levels, and enhanced estrogen signaling, in PAH patients. Evidence suggests that exuberant estrogen signaling causes a perturbation of mitochondrial function and energy substrate utilization in both sexes. However, systemic estrogen level elevation is not uniform among patients, and the affinity of the pulmonary vascular bed for estrogens is unknown. In preliminary studies of prevalent PAH patients, estradiol (E2) levels dropped across the pulmonary vasculature suggestive of E2 uptake by the lungs; those patients with a high transpulmonary gradient (pre- minus post-capillary) had a higher mean pulmonary artery pressure at diagnosis.

Investigators previously confirmed that urine 16α-hydroxyestrone (16αOHE1) is elevated at least 2-fold in females and males with PAH, consistent with data from other groups that estrogens are elevated in PAH. 16αOHE1 is an estrogen metabolite with high affinity for the canonical estrogen receptors (ESRα and ESRβ) and thus an active estrogen. Investigators published that in a transgenic mouse model of PAH, administration of 16αOHE1 significantly increased PAH penetrance concomitant with features of oxidant stress including elevated isoprostanes (IsoPs) and isofurans (IsoFs). Those animals also developed insulin resistance and mitochondrial dysfunction, characteristics investigators have described during the current PPG in humans with PAH. Concomitantly, through ESR signaling, 16αOHE1 reduced PPARγ expression via reduction in PGC1α. By co-administering drugs to block extra-gonadal estrogen synthesis and receptor signaling investigators were able to prevent or reverse the cellular metabolic defects and pulmonary vascular phenotype in investigators' transgenic model system.

The capacity for enhanced estrogen signaling, represented by elevated blood E2 levels, elevated urinary 16αOHE1, and specific genetic variants, is a characteristic of PAH patients of both sexes in several studies. Experimental data from investigators' group and others support the concept that estrogen antagonism may be beneficial for humans with PAH. However, investigators recognize that not all subjects will benefit from estrogen antagonism, making a 'one size fits all' approach too narrow.

Investigators and others have shown that estrogens directly alter pulmonary vascular cell homeostasis and gene expression, including reduction in BMPR2 expression and signaling via ESR; and, experimental PAH models demonstrate increased expression of aromatase, an enzyme which converts androgens to estrogens, in the lungs. But no human studies investigate the direct contribution of the pulmonary circulation to estrogen avidity, ESR density, and outcomes. Investigators propose to evaluate the influence of estrogens on the pulmonary vasculature and cardiac function, using incident and prevalent PAH cases to reduce confounding by disease course. Findings from this study should help determine patients most likely to have a beneficial response to estrogen antagonism, supporting the overall project goal to improve "precision medicine" approaches in PAH.

Investigators hypothesize that blood-based and radiologic markers of estrogen burden will support the determination of a phenotype profile of subjects with PAH for whom estrogen antagonism will be an effective therapeutic approach. In a cohort of PAH patients, investigators will determine if transpulmonary (change pre- to post-pulmonary capillary bed) E2 levels and/or lung ESR density associate with disease severity at cardiac catheterization, functional capacity, time to clinical worsening, and oxidant stress.

Specific Aim 1: To test the hypothesis that among PAH patients, transpulmonary (TP) E2 gradient associates with a more severe hemodynamic profile and worse 1 year outcomes.

Specific Aim 2: To test the hypothesis that among PAH patients, higher lung ESR density associates with a more severe hemodynamic profile and worse 1 year outcomes.

These studies may ultimately lead to novel discoveries in the transpulmonary gradient of sex hormones, investigate a novel imaging approach in PAH, optimize the ability to precisely determine the correct patient for sex hormone modification, and potentially support the development of novel therapeutic targets in PAH. The data collected in this study will also synergize with an ongoing NIH-supported clinical trial to investigate the use of sex hormone modification as a therapeutic approach for PAH:

ClinicalTrials.gov Identifier: NCT03528902.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 years or older
* Group 1: PH Patients, who have precapillary PH (PAH). Patients with and without a known PAH-associated gene mutation (e.g., a BMPR2 mutation) (i.e. those with HPAH and those with IPAH) will be identified based on previous genotyping. Investigators define pulmonary hypertension diagnostically by accepted clinical and cardiac catheterization criteria, including mean pulmonary arterial pressure of more than 25 mmHg. Precapillary PH (PAH) cases have pulmonary capillary or left atrial pressure of ≤15 mm Hg, and exclusion of other causes of pulmonary hypertension in accordance with accepted international standards of diagnostic criteria.
* Group 2: PVH Patients, who have pulmonary hypertension secondary to left heart disease. PVH cases have left ventricular (LV) filling pressure >15 mmHg (measured by the pulmonary artery occlusion pressure or left ventricular end-diastolic pressure) and a diastolic pressure gradient <7mmHg, indicating the absence of pulmonary vascular disease. Inclusion in this group will require a clinical diagnosis of systolic or diastolic heart failure and right heart catheterization on at least one occasion demonstrating elevated pulmonary wedge pressure and a normal (< 16mmHg) trans-pulmonary gradient
* Group 3: Healthy Control Patients, who have no known history of cardiopulmonary disease recruited from the Vanderbilt Research Notification Distribution List and the population at large.

Exclusion Criteria:

1. Subjects with the following concurrent diagnoses

   * Type 1 Diabetes Mellitus
   * Polycystic ovarian disease
   * Breast/uterine/endometrial cancer
2. Subjects with the following concurrent exposures

   * Use of hormone modifying therapy
   * Use of hormone-containing pharmaceuticals including hormone replacement therapy.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group 1 pulmonary hypertension (PAH) patients compared to Group 2 PH (pulmonary venous hypertension, PVH) patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
To correlate lung ESR density with pulmonary vascular resistance (PVR) | Day 1
  Positron emission tomography (PET) with ESR-targeting radiopharmaceuticals is a noninvasive method for assessing regional ESR expression in vivo. For example, multiple studies have shown that the detection of ESR positive tissue by 18F-FES PET is reliable and that 18F-FES uptake correlates well with immunohistochemical scoring for ESR density. We will determine the relationship, if any, between the density of ESR in the lungs of subjects, and pulmonary vascular resistance (PVR), measured in Woods Units, acquired at time of recent cardiac catheterization.

SECONDARY OUTCOMES:
Survival at one year | 1 year
  We will determine the association of lung ESR density with survival within one year of the PET scan study.

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Austin, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Vanderbilt may share subject information, without identifiers, to others or use it for other research projects not listed in the consent form. Vanderbilt, Dr. Eric Austin, and his staff will comply with any and all laws regarding the privacy of such information. There are no plans to pay subjects for the use or transfer of this de-identified information.
  All efforts, within reason, will be made to keep subjects protected health information (PHI) private. All federal privacy laws will be followed.
  As part of the study, Dr. Austin and his study team may share the results of subject's study blood work, PET CT, and catheterization data as well as parts of their medical record in de-identified manner. The Federal Government Office for Human Research Protections and the Vanderbilt University Institutional Review Board might review this study to ensure investigators are following all local and Federal guidelines for patient protection.

DOCUMENTS (1):
  • Informed Consent Form (2022-09-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT04280523/ICF_000.pdf